CLINICAL TRIAL: NCT03272932
Title: A Cross-sectional Study to Assess the Proportion and Clinical Characteristics of Asthma and COPD Overlap for Patients With Asthma and COPD in Hong Kong.
Brief Title: Clinical Characteristics of Asthma and COPD Overlap for Patients With Asthma and COPD in Hong Kong
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fanny W.S. Ko, Honorary Clinical Associate Professor, Chinese University of Hong Kong
Other Study IDs: CCUHK_Resp_ACOS_v1(5Apr2017)
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: COPD; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be stored for future genetic studies. As there is currently no good biomarker or genetic tests that can identify the cause or suggest the diagnosis of Asthma COPD overlap, this study would like to explore into this.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study is to assess the prevalence of Asthma COPD Overlap in subjects with diagnosed asthma and chronic obstructive pulmonary disease (COPD). The subsequent morbidity and mortality of subjects will be followed up for 3 years.

DETAILED DESCRIPTION:
Rationale:

Around 15 to 20% of COPD patients have features of asthma. These patients have more frequent and more severe exacerbations, and higher medical utilization. The Global Initiative for Asthma (GINA) and Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines have given joint recommendations on the identification, diagnosis and treatment of these patients having Asthma-COPD Overlap (ACO). These are at present expert opinions and further studies are needed to establish the optimal definitions and treatment options. The recommendations proposed by the guidelines have been adapted for use in the Asia area countries. Nonetheless, the application to clinical practice has not been well established and there are no prevalence data available on the COPD with asthma symptom population or asthma with COPD symptoms population based on the recommended features for identification. This is the current data gap in Asia.

Primary objective:

To determine the proportion and clinical characteristics of patients with ACO as defined by the joint GINA and GOLD recommendation amongst diagnosed COPD and asthma patients seen at the out-patient clinics

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfil all of the following criteria:

* All patients with confirmed diagnosis of COPD (post-bronchodilator FEV1/FVC<0.7 based on the medical records) 1 or asthma (defined as those with a consistent history and prior documented evidence of variable airflow obstruction, with evidence of an increase in FEV1 greater than 12% or 400 mL following bronchodilator or bronchial hyperresponsiveness on bronchial provocation testing, when stable) 6
* Aged >40 years old
* Signed written informed consent to participate in the study

Exclusion Criteria:

* Patients currently with acute exacerbation of COPD by GOLD definition (any worsening of a patient's respiratory symptoms that is beyond normal day-to-day variations and requires a change in medication) 1 or acute exacerbation of asthma by GINA guideline. 6
* Patients with respiratory diseases that can show similar symptoms to chronic airway diseases such as bronchiectasis, tuberculosis (TB)-destroyed lung parenchyma, endobronchial TB, and lung cancer, or those who have history of these diseases based on physician's judgment
* Patients currently diagnosed with pneumonia and acute bronchitis
* Patients currently randomized in other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with asthma or COPD
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of prevalence of Asthma COPD overlap among the asthma and COPD subjects. | 3 years
  To determine the proportion and clinical characteristics of patients with ACO as defined by the joint GINA and GOLD recommendation amongst diagnosed COPD and asthma patients seen at the out-patient clinics. (Assessment: % of subjects with ACO among patients with asthma and COPD respectively)

SECONDARY OUTCOMES:
Percentage of patient with treatment that is different from the guidelines recommendation | 3 years
  To evaluate the gap between guideline recommendations and real-world clinical practice in identifying COPD patients with asthma and asthma patients with COPD
The percentages of patients on various medications (e.g. inhaled steroid, LABA, LAMA) | 3 years
  To review the medications given to COPD patients with asthma and asthma patients with COPD compared to guideline recommendations
The pecentages of patients receiving different symptoms control assessments (e.g. use of Asthma control test, use of COPD assessment test) | 3 years
  To review the current practices of symptom control assessment
Percentages of subjects with morbidity (e.g. congestive heart failure) | 3 years
  To assess the 3 year morbidity of ACO patient compared to COPD and asthma patients.
Percentages of subjects with mortality | 3 years
  To assess the 3 year mortality of ACO patient compared to COPD and asthma
Percentages of patients with various Genetic markers | 3 years
  Genetic markers got differentiating ACO patients from patients with COPD or asthma

CONTACTS AND LOCATIONS:
Overall Officials: Fanny Ko, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No